CLINICAL TRIAL: NCT00419055
Title: Outpatient Percutaneous Coronary Intervention in a Selected, Stable Patient Population
Brief Title: Outpatient Percutaneous Coronary Intervention
Status: Terminated | Type: Observational
Why Stopped: Stopped early due to inability to recruit full 100 subjects over 2 years
Sponsor: University of Pennsylvania (Other)
Collaborators: Abbott Medical Devices (Industry); The Medicines Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 801441
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Coronary Artery Disease
Keywords: percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1 Control: Patients are discharged the day after PCI
  Interventions: Procedure: Early discharge after percutaneous coronary intervenntion
- 2 Study group: Patients will be discharged 4-6 hrs after PCI
  Interventions: Procedure: Early discharge after percutaneous coronary intervenntion

INTERVENTIONS:
Procedure: Early discharge after percutaneous coronary intervenntion — Eligible patients receive Bivalirudin at the standard dose during PCI and all have to be eligible for femoral access seal.

SUMMARY:
To determine the safety and feasibility of same day discharge after elective coronary percutaneous intervention in a selected stable patient population. The hypothesis to be tested is that in an appropriately selected stable coronary artery disease population post percutaneous coronary intervention, early discharge is safe and feasible.

DETAILED DESCRIPTION:
A select stable population of patients undergoing percutaneous coronary intervention are randomized to standard of care in-hospital stay for one night or early discharge to a nearby hotel. During PCI, patients receive bivalirudin as their anti-coagulant and also must be eligible for an angioseal closure device. Patients that stay overnight in the hotel must be accompanied by a family member. They return to the cath lab the next day for groin check and blood work. Satisfaction questionnaires are filled out by all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable coronary artery disease scheduled for elective percutaneous coronary intervention

Exclusion Criteria:

* Patients with acute coronary syndrome, patients with an MI within 30 days, an ejection fraction <30%, those with history of IV Dye allergy, creatinine level>2.2, those with increased risk of infection, those with history of bleeding diathesis or anemia (hemoglobin<11.0 g/dl, platelets <100,000 tho/ul)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients less than 75 years who have undergone PCI
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2004-08; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoints are patient satisfaction and safety. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Howard C Herrmann, M.D., Principal Investigator — University of Pennsylvania; Ruchira Glaser, M.D., Principal Investigator — University of Pennsylvania